CLINICAL TRIAL: NCT07198230
Title: Drug-Eluting Bead-Based Transarterial Chemoembolization (DEB-TACE) as a Local Salvage Therapy for Large Lesions in Relapsed and Refractory Diffuse Large B-Cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Ting YANG (Other)
Responsible Party: Sponsor-Investigator, Ting YANG, Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: DLBCL-DEBTACE-01
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Large B-Cell Lymphoma; Relapsed and Refractory; Transarterial Chemoembolization
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DEB-TACE: Drug-Eluting Bead-Based Transarterial Chemoembolization (DEB-TACE) as a Salvage Therapy for Recurrent and Refractory Diffuse Large B-Cell Lymphoma with Bulky Lesions

SUMMARY:
Current exploration of local therapies for large Diffuse Large B-Cell Lymphoma (DLBCL) masses remains in its infancy. This study aims to retrospectively evaluate the safety, efficacy, and tolerability of Drug-Eluting Bead-Based Transarterial Chemoembolization (DEB-TACE) for treating recurrent and refractory DLBCL masses. It seeks to establish a novel local salvage treatment strategy for such patients while providing preliminary theoretical foundations and clinical data to support future large-scale, multicenter clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18 to 75 years; (2) Pathologically confirmed diffuse large B-cell lymphoma (DLBCL); (3) Recurrence or treatment resistance following multiple therapeutic regimens (e.g., chemotherapy, immunotherapy, targeted therapy), with at least one clearly defined bulky lesion (maximum diameter ≥5 cm or imaging evidence of bulky lesion); (4) Imaging studies (CT, MRI, or PET-CT) confirm rich blood supply to the lesion, making it suitable for transarterial interventional therapy; (5) History of favorable response to doxorubicin-based agents during prior systemic therapy; (6) ECOG performance status ≤ 2; (7) Blood counts, hepatic and renal function, and coagulation parameters meet the following criteria:

  * Platelet count ≥ 30 × 10^9/L;
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the ULN;
  * Serum creatinine ≤ 2.5 times the upper limit of normal (ULN);
  * Prothrombin time international normalized ratio (INR) ≤ 1.5. (8) The patient has previously undergone at least one DEB-TACE treatment at this institution.

Exclusion Criteria:

* (1) Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction, or other serious comorbidities rendering them unable to tolerate interventional therapy; (2) Patients with active or uncontrolled severe infections; (3) Patients with severe coagulation disorders or bleeding tendencies; (4) Pregnant or lactating women, or patients planning pregnancy during the study period; (5) Allergy or contraindications to drug-eluting microsphere materials or chemotherapy drugs; (6) Psychiatric disorders or cognitive impairment preventing treatment compliance and follow-up; (7) Other conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed and refractory diffuse large B-cell lymphoma with bulky lesions
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 months
  The objective response rate (ORR) refers to the proportion of patients whose tumor volume reduction reaches a predetermined threshold and is maintained for the minimum required duration. It is calculated as the sum of complete response (CR) and partial response (PR) rates, i.e., ORR = CR + PR.
Local Response Rate | 3 months
  The local lesion response rate typically refers to the proportion of local lesions that show a reduction in volume or improvement in symptoms following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided